CLINICAL TRIAL: NCT00757029
Title: Association Between Norepinephrine Transporter Polymorphism and Response of Methylphenidate
Brief Title: Pharmacogenetic Study of Methylphenidate in Attention Deficit/Hyperactivity Disorder(ADHD)
Acronym: NETADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NETADHD
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2010-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Methylphenidate; Pharmacogenetics
Keywords: ADHD,; norepinephrine transporter; pharmacogenetics
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Time; Norepinephrine Plasma Membrane Transport Proteins; Polymorphism, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Other)
  Interventions: Genetic: norepinephrine transporter polymorphism,

INTERVENTIONS:
Genetic: norepinephrine transporter polymorphism, — OROS methylphenidate (Concerta) monopharmacotherapy dose : 18-54mg duration : 8 weeks genotyping : norepinephrine transporter (SLC6A2) polymorphism
  Other Names: OROS methylphenidate (Concerta) monopharmacotherapy; dose : 18-54mg; duration : 8 weeks; genotyping : norepinephrine transporter (SLC6A2) polymorphism

SUMMARY:
The noradrenergic system plays a known role in attentional systems and suspected causal role in attention deficit/hyperactivity disorder(ADHD).Methylphenidate also has been suspected as a inhibitor of norepinephrine transporter(SLC6A2). The investigators hypothesis is that norepinephrine transporter polymorphism is associated with responses and adverse effects of OROS-methylphenidate in treatment of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* ADHD
* Physically healthy

Exclusion Criteria:

* Neurological illness
* Concurrent additional psychiatric treatment
* < IQ 70
* Psychotic disorder
* Major mood disorder needed other psychiatric medication
* Significant suicidal ideation
* Pervasive developmental disorder

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Korean ADHD Rating scale-parent version (KARS) | baseline,1,2,4,8 weeks

SECONDARY OUTCOMES:
Barkely side effect rating scale | 1,2,4,8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea